CLINICAL TRIAL: NCT00005289
Title: Risk Factors in Bronchopulmonary Dysplasia (Newborn Lung Project)
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1997-152; R01HL038149 (NIH); 1997-152 (Other: Institutional Review Board); 2002-209 (Other: Institutional Review Board)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Bronchopulmonary Dysplasia; Lung Diseases; Respiratory Distress Syndrome
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Lung Diseases; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1988-1991
- 2003-2004

SUMMARY:
To investigate risk factors in bronchopulmonary dysplasia (BPD) and to elucidate the relationship between BPD, acute lung disease severity, respiration-related variables, water balance, nutrition, familial predisposition, and environmental, pregnancy, and delivery parameters.

DETAILED DESCRIPTION:
BACKGROUND:

Despite many improvements in neonatal intensive care during the decade from 1977 to 1987, infant respiratory distress syndrome remained a major public health problem. Increasing survival among premature infants led to the emergence of BPD as the major chronic respiratory disorder of infancy. The vast majority of BPD occurs in very low birth weight infants weighing less than 1,500 grams.

Although the incidence of low birth weight births declined from 1977 to 1987, the rate of very low birth weight births remained unchanged. These infants had a relative risk of neonatal death almost 200 times greater than full-term infants. Among survivors, eight percent had evidence of chronic pulmonary disease at forty weeks of age. The Institute of Medicine reported that very low birth weight infants who survived to one year of age were hospitalized for an average of 57 days after birth versus 3.5 days for full-term infants. Up to forty percent of these infants would be re-hospitalized almost two times for an average of 16 days versus 8.7 percent of normal birth weight infants for an average of 8 days.

DESIGN NARRATIVE:

The study had a nested case-control design. In the first year of the project, the diagnosis of BPD was standardized and a scoring system developed for grading the severity of the disease. Baseline data were collected on very low birth weight neonates admitted to seven participating neonatal intensive care units. Maternal interviews were conducted for neonates surviving seven days. The purpose of the interview was to collect information which m;ight be related to a predisposition to BPD, respiratory distress syndrome, or prematurity. Specific areas addressed included familial diseases in general and respiratory diseases in particular, familial patterns of prematurity, pregnancy and birth history, circumstances surrounding delivery, environmental exposures, health habits such as smoking, and socioeconomic variables. Severity scoring and diagnosis of the infants were based on the hospital log and routine x-rays. Final analysis compared infants with BPD to those without BPD, controlling for confounders and placing special emphasis on interaction effects. Full-term neonates served as controls.

The study was renewed in 1994 in order to re-contact at age 4-5, an existing cohort of 634 children with birth weight below 1501 grams. This cohort was unique in being representative of all very low birth weight survivors in a geographic area, and in being born during a time period of rapid advances in neonatal care (Aug 1, 1988-June 30, 1991). These children were enrolled at admission to any of 6 neonatal intensive care units (NlCUs) in Wisconsin and Iowa, and had extensive data already collected. The re-contact consisted of a telephone interview with parents, including standardized functional assessment. Information on health care and major diagnoses was also collected and verified by medical record abstracting. Information on socioeconomic and insurance status was obtained. The study responded to a need for global assessment of very low birth weight survivors, since most previous studies in the United States focused on specific morbidity outcomes. Special features of already existing data included scoring of respiratory distress syndrome and bronchopulmonary dysplasia severity with new validated severity indices, baseline family health history information and perinatal data. The cohort also spanned the time period from before general availability of exogenous surfactant to its availability as an investigational new drug (8/1/89) and availability for marketing (8/1/90). The study therefore provided an opportunity to investigate the long term effectiveness of this new therapy in an unselected NlCU population. The data were analyzed to describe the overall status of the cohort, to examine trends in outcomes across the time period, to find predictors of outcome among the neonatal and socioeconomic indicators and to investigate whether there was variability between centers.

The study was renewed in 1998 to continue follow-up of the cohort of 403 very low birth weight neonatal care survivors, born during August 1988-June1991. The time period of birth includes the approval dates for surfactant therapy. Hence, the first children to be treated with surfactant in general neonatal intensive care units (NICU) are now entering school age, providing an opportunity to evaluate school performance and to assess true chronicity of respiratory limitations. A large NICU and follow-up data base on the cohort contains extensive baseline assessment of respiratory disease, neonatal treatments and diagnoses, as well as functional assessment, health status and health care utilization at ages 4-6. The addition of data up to age 10 will confirm or dispute findings that functional outcome may be lower among children born after surfactant was released for marketing, and that the prevalence of long-term respiratory problems has remained the same. The new outcome data to be collected include school performance from school records and parent and teacher questionnaires, respiratory function by peak flow meters and respiratory symptoms and medications by parent interviews and questionnaires.

The study was renewed in 2002 to continue research in the evolving risk factors and outcomes of bronchopulmonary dysplasia (BPD) and other neonatal conditions of very low birth weight (VLBW, < 1500g) infants and children. The renewal will comprehensively document the neonatal and early childhood course and outcomes of all VLBW births in Wisconsin occurring during the calendar years 2003 and 2004 (800-850 per year), using established methodology with added risk factor information to examine currently proposed inflammatory hypotheses of BPD etiology. The study will also implement and validate new diagnostic criteria for the severity of BPD developed by a recent NIH workshop.

ELIGIBILITY:
- Birthweight less than 1500 grams

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2202 (Actual)
Dates: Start 1987-07; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mari Palta — University of Wisconsin, Madison

REFERENCES:
- [Background] Farrell ET, Bates ML, Pegelow DF, Palta M, Eickhoff JC, O'Brien MJ, Eldridge MW. Pulmonary Gas Exchange and Exercise Capacity in Adults Born Preterm. Ann Am Thorac Soc. 2015 Aug;12(8):1130-7. doi: 10.1513/AnnalsATS.201410-470OC. PMID 26053283
- [Result] Palta M, Gabbert D, Fryback D, Widjaja I, Peters ME, Farrell P, Johnson J. Development and validation of an index for scoring baseline respiratory disease in the very low birth weight neonate. Severity Index Development and Validation Panels and Newborn Lung Project. Pediatrics. 1990 Nov;86(5):714-21. PMID 2235225
- [Result] Palta M, Gabbert D, Weinstein MR, Peters ME. Multivariate assessment of traditional risk factors for chronic lung disease in very low birth weight neonates. The Newborn Lung Project. J Pediatr. 1991 Aug;119(2):285-92. doi: 10.1016/s0022-3476(05)80746-2. PMID 1861218
- [Result] Palta M, Weinstein MR, McGuinness G, Gabbert D, Brady W, Peters ME. A population study. Mortality and morbidity after availability of surfactant therapy. Newborn Lung Project. Arch Pediatr Adolesc Med. 1994 Dec;148(12):1295-301. doi: 10.1001/archpedi.1994.02170120057009. PMID 7951809
- [Result] Palta M, Sadek-Badawi M, Evans M, Weinstein MR, McGuinnes G. Functional assessment of a multicenter very low-birth-weight cohort at age 5 years. Newborn Lung Project. Arch Pediatr Adolesc Med. 2000 Jan;154(1):23-30. PMID 10632246
- [Result] Evans M, Palta M, Sadek M, Weinstein MR, Peters ME. Associations between family history of asthma, bronchopulmonary dysplasia, and childhood asthma in very low birth weight children. Am J Epidemiol. 1998 Sep 1;148(5):460-6. doi: 10.1093/oxfordjournals.aje.a009671. PMID 9737558
- [Result] Palta M, Sadek M, Lim TS, Evans M, McGuinness G. Association of tocolytic therapy with antenatal steroid administration and infant outcomes. Newborn Lung Project. Am J Perinatol. 1998 Feb;15(2):87-92. doi: 10.1055/s-2007-993904. PMID 9514131
- [Result] Palta M, Sadek M, Barnet JH, Evans M, Weinstein MR, McGuinness G, Peters ME, Gabbert D, Fryback D, Farrell P. Evaluation of criteria for chronic lung disease in surviving very low birth weight infants. Newborn Lung Project. J Pediatr. 1998 Jan;132(1):57-63. doi: 10.1016/s0022-3476(98)70485-8. PMID 9470001
- [Result] Palta M, Sadek M, Gabbert D, Brady W, Weinstein MR, McGuinness G, Peters ME. The relation of maternal complications to outcomes in very low birthweight infants in an era of changing neonatal care. Am J Perinatol. 1996 Feb;13(2):109-14. doi: 10.1055/s-2007-994303. PMID 8672182
- [Result] Weinstein MR, Peters ME, Sadek M, Palta M. A new radiographic scoring system for bronchopulmonary dysplasia. Newborn Lung Project. Pediatr Pulmonol. 1994 Nov;18(5):284-9. doi: 10.1002/ppul.1950180504. PMID 7898966
- [Result] Palta M, Sadek-Badawi M, Sheehy M, Albanese A, Weinstein M, McGuinness G, Peters ME. Respiratory symptoms at age 8 years in a cohort of very low birth weight children. Am J Epidemiol. 2001 Sep 15;154(6):521-9. doi: 10.1093/aje/154.6.521. PMID 11549557
- [Result] Hagen EW, Palta M, Albanese A, Sadek-Badawi M. School achievement in a regional cohort of children born very low birthweight. J Dev Behav Pediatr. 2006 Apr;27(2):112-20. doi: 10.1097/00004703-200604000-00005. PMID 16682874
- [Result] Palta M, Sadek-Badawi M, Madden K, Green C. Pulmonary testing using peak flow meters of very low birth weight children born in the perisurfactant era and school controls at age 10 years. Pediatr Pulmonol. 2007 Sep;42(9):819-28. doi: 10.1002/ppul.20662. PMID 17659600
- [Result] Hagen EW, Sadek-Badawi M, Albanese A, Palta M. A comparison of Wisconsin neonatal intensive care units with national data on outcomes and practices. WMJ. 2008 Nov;107(7):320-6. PMID 19180870
- [Result] Hagen EW, Sadek-Badawi M, Carlton DP, Palta M. Permissive hypercapnia and risk for brain injury and developmental impairment. Pediatrics. 2008 Sep;122(3):e583-9. doi: 10.1542/peds.2008-1016. PMID 18762492
- [Result] Palta M, Sadek-Badawi M, Carlton DP. Association of BPD and IVH with early neutrophil and white counts in VLBW neonates with gestational age <32 weeks. J Perinatol. 2008 Sep;28(9):604-10. doi: 10.1038/jp.2008.65. Epub 2008 Jun 19. PMID 18563166
- [Result] Palta M, Sadek-Badawi M. PedsQL relates to function and behavior in very low and normal birth weight 2- and 3-year-olds from a regional cohort. Qual Life Res. 2008 Jun;17(5):691-700. doi: 10.1007/s11136-008-9346-1. Epub 2008 May 6. PMID 18459069
- [Result] Hagen EW, Sadek-Badawi M, Palta M. Daycare attendance and risk for respiratory morbidity among young very low birth weight children. Pediatr Pulmonol. 2009 Nov;44(11):1093-9. doi: 10.1002/ppul.21104. PMID 19824048
- [Result] McManus BM, Robert SA, Albanese A, Sadek-Badawi M, Palta M. Racial disparities in health-related quality of life in a cohort of very low birthweight 2- and 3-year-olds with and without cerebral palsy. Dev Med Child Neurol. 2011 May;53(5):467-9. doi: 10.1111/j.1469-8749.2011.03923.x. Epub 2011 Mar 17. PMID 21410692
- [Result] McManus BM, Robert SA, Albanese A, Sadek-Badawi M, Palta M. Relationship between neighborhood disadvantage and social function of Wisconsin 2- and 3-year-olds born at very low birth weight. Arch Pediatr Adolesc Med. 2011 Feb;165(2):119-25. doi: 10.1001/archpediatrics.2010.185. Epub 2010 Oct 4. PMID 20921342
- [Result] Witt WP, Litzelman K, Spear HA, Wisk LE, Levin N, McManus BM, Palta M. Health-related quality of life of mothers of very low birth weight children at the age of five: results from the Newborn Lung Project Statewide Cohort Study. Qual Life Res. 2012 Nov;21(9):1565-76. doi: 10.1007/s11136-011-0069-3. Epub 2011 Dec 10. PMID 22161725
- [Result] McManus BM, Robert S, Albanese A, Sadek-Badawi M, Palta M. Racial disparities in health-related quality of life in a cohort of very-low-birth-weight 2- and 3-year-olds with and without asthma. J Epidemiol Community Health. 2012 Jul;66(7):579-85. doi: 10.1136/jech.2010.132886. Epub 2011 Feb 17. PMID 21330462
- [Result] Bates ML, Pillers DA, Palta M, Farrell ET, Eldridge MW. Ventilatory control in infants, children, and adults with bronchopulmonary dysplasia. Respir Physiol Neurobiol. 2013 Nov 1;189(2):329-37. doi: 10.1016/j.resp.2013.07.015. Epub 2013 Jul 22. PMID 23886637
- [Result] McManus BM, Robert S, Albanese A, Sadek-Badawi M, Palta M. Predictors of receiving therapy among very low birth weight 2-year olds eligible for Part C early intervention in Wisconsin. BMC Pediatr. 2013 Jul 11;13:106. doi: 10.1186/1471-2431-13-106. PMID 23845161
- [Result] Haraldsdottir K, Watson AM, Goss KN, Beshish AG, Pegelow DF, Palta M, Tetri LH, Barton GP, Brix MD, Centanni RM, Eldridge MW. Impaired autonomic function in adolescents born preterm. Physiol Rep. 2018 Mar;6(6):e13620. doi: 10.14814/phy2.13620. PMID 29595875
- [Result] Bates ML, Farrell ET, Eldridge MW. Abnormal ventilatory responses in adults born prematurely. N Engl J Med. 2014 Feb 6;370(6):584-5. doi: 10.1056/NEJMc1311092. No abstract available. PMID 24499235
- [Result] Goss KN, Beshish AG, Barton GP, Haraldsdottir K, Levin TS, Tetri LH, Battiola TJ, Mulchrone AM, Pegelow DF, Palta M, Lamers LJ, Watson AM, Chesler NC, Eldridge MW. Early Pulmonary Vascular Disease in Young Adults Born Preterm. Am J Respir Crit Care Med. 2018 Dec 15;198(12):1549-1558. doi: 10.1164/rccm.201710-2016OC. PMID 29944842